CLINICAL TRIAL: NCT04835987
Title: Prospective Monocentric Evaluation of the Autonomic Nervous System in Patients Undergoing Esophagectomy for Cancer
Brief Title: Evaluation of the Autonomic Nervous System in Patients Undergoing Esophagectomy for Cancer
Acronym: PROSNACO
Status: Withdrawn | Type: Observational
Why Stopped: Due to a lack of staff in the department, no inclusion could be realized.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH250; 2020-A03326-33 (Other: ANSM)
Record Dates: First submitted 2021-03-26; First posted 2021-04-08 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; surgery; Holter-ECG
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Holter ECG — Measurement of the modification of the sympathomimetic balance
Behavioral: Questionary — Lifestyle questionary (time spent in front of television, physical activity)
Diagnostic Test: Pupillometry — Monitoring of nociception and autonomic nervous system by pupillometry in intraoperative.

SUMMARY:
Esophageal surgery is a complex surgery, with high post-operative morbidity and mortality. The incidence of complications associated with esophagectomy varies from 17% to 74%, in the literature. A section of vagus nerves is conventionally performed during esophagectomy for cancer, because of oncological margins. The vagus nerve is responsible for the parasympathetic innervation at the gastrointestinal level, but also at the cardiac and pulmonary level. The post-operative morbidity of these procedures could be linked in part to the bilateral section of the vagus nerves, because of their impact on the autonomous regulation of this vital functions. The main objective of the study is to find a modification of the sympathomimetic balance pre and post operatively, in patients undergoing esophagectomy.

DETAILED DESCRIPTION:
The sympathomimetic balance was measured using a Holter-ECG heart rate monitor. The parameters collected were used to calculate the variability of the heart rate, the high frequencies (HF, reflection of the parasympathetic system), the low frequencies (LF, reflection of the sympathetic system and the parasympathetic system) and the ratio // LF / HF (reflection of the sympathetic activity) thanks to Fourier analysis and the use of HRVanalysis software.

The measurements were taken at night, to overcome the great sympathomimetic variabilities due to external stimulations during the day: one night 3 month before surgery/before the first chemotherapy, one night between 2 and 4 weeks before hospitalization (remotely of possible chemotherapy), the night before the intervention (context of hospitalization and preoperative stress), one night between D7 and D10 (context of hospitalization, and distance from anesthetic drugs), one night at home between 4 and 8 weeks post-operative, and one night at home at 3 months post-operative.

The measurements were therefore not carried out the first nights following the intervention to overcome the anesthetic drugs that affect the balance of the autonomic nervous system.

A baroreflex measurement was carried out at the patient's entrance, the day before the intervention, during hospitalization, and the day of discharge. This measure was renewed at 3 months.

A measurement of patient activity was carried out preoperatively by wearing an actimeter watch for 1 week then renewed at 3 months.

A Respiratory Functional Exploration associated with a stress test with calculation of the VO2max is systematically carried out before the esophageal surgery. A Respiratory Functional Exploration was renewed 4 to 8 weeks after the intervention, and then at 3 months. the 6-minute walk test was performed at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Esophagectomy for cancer
* written and oral agreement

Exclusion Criteria:

* pregnant women,
* patients with permanent atrial fibrillation,
* patients with pace-maker
* Patients under guardianship/curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population aged over 18 years with esophagectomy for cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of Standard deviation of all NN (SDNN) (ms) | before surgery
  Analysis of Standard deviation of all NN (SDNN) intervals, over the entire registration period, provides information on global variability. Measured by Holter results. Day 0 = surgery
Analysis of Standard deviation of all NN (SDNN) (ms) | day 7 to day 90
  Analysis of Standard deviation of all NN (SDNN) intervals, over the entire registration period, provides information on global variability. Measured by Holter results. Day 0 = surgery

SECONDARY OUTCOMES:
HF activity | before surgery : Day -82, Day -30, Day -1
  Day 0 = surgery measured with the Holter Electrocardiogram
LF activity | before surgery : Day -82, Day -30, Day -1
  Day 0 = surgery measured with the Holter Electrocardiogram
LF/HF ratio | before surgery : Day -82, Day -30, Day -1
  Day 0 = surgery measured with the Holter Electrocardiogram
HF activity | after surgery : day 7, day 60, day 90
  Day 0 = surgery measured with the Holter Electrocardiogram
LF activity | after surgery : day 7, day 60, day 90
  Day 0 = surgery measured with the Holter Electrocardiogram
LF/HF ratio | after surgery : day 7, day 60, day 90
  Day 0 = surgery measured with the Holter Electrocardiogram
change in baroreflex | Day -1, Day 7, day discharge, day 90
  baroreflex sensitivity : ms/mmHg Day 0 = surgery
modify the respiratory functional exploration | Day -30, Day 30, Day 60
  Peak expiratory volume per second : L Day 0 = surgery
intraoperative pupillometry | during surgery
  pupillary diameter : mm
physical capacity | Day-30, Day 30, Day 90
  walking distance in 6 minutes Day 0 = surgery

CONTACTS AND LOCATIONS:
Overall Officials: EVE HUART, MD, Principal Investigator — CHU ST ETIENNE
Locations (1):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No